CLINICAL TRIAL: NCT03979963
Title: Depressive Symptoms and Emotion Regulation Following Outpatient Cognitive Behavioral Therapy for Depression: a Longitudinal Study
Brief Title: Depressive Symptoms and Emotion Regulation Following Cognitive Behavioral Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Verena Zimmermann, Research Associate, Heidelberg University
Other Study IDs: Depression & ER
Record Dates: First submitted 2019-05-27; First posted 2019-06-10 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Depression
Keywords: Depression; Emotion Regulation; Cognitive Behavioral Therapy; Ecological Momentary Assessment
MeSH Terms: conditions — Depression; Emotional Regulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates depressive symptoms and the use of emotion regulation strategies over the course of a two-year period in participants terminating outpatient cognitive behavioral therapy for depression. The main objective of the study is to examine if changes in the use of certain emotion regulation strategies (e.g. reappraisal, rumination) predict depression relapse or changes in depressive symptoms after the completion of outpatient cognitive behavioral therapy.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years
* regular termination of outpatient cognitive behavioral therapy for depression (or premature termination agreed upon by both the therapist and the patient because of symptom improvement after at least 12 sessions)
* last therapy session not more than two weeks prior to enrollment
* self-reported improvement in depressive symptoms as a result of cognitive behavioral therapy
* possession of a smartphone (operating system: Android or iOS) with Internet access
* possession of a laptop/desktop computer with Internet access
* familiarity with apps and the Internet
* fluency in German language

Exclusion Criteria:

* premature termination of outpatient cognitive behavioral therapy (exception: termination agreed upon by both the therapist and the patient because of symptom improvement)
* BDI-II score ≥ 20
* acute substance use disorder (< 3 months)
* current or past psychotic disorder
* current or past (hypo)manic episode
* acute suicidality
* severe neurological disorder/cerebral damage
* severe physical/medical illness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have recently completed outpatient cognitive behavioral therapy for depression
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in ecological momentary assessment scores | 0, 3, 6, 9, 12, 15, 18, 21, and 24 months after completion of cognitive behavioral therapy
  Change in ecological momentary assessment scores. Data will be collected using the smartphone app EmoTrack2. The app measures emotions experienced, context factors of the emotional experiences, and emotions regulation strategies used (five measurements per day over a period of seven consecutive days).
Change in the mental disorders diagnosed with the Structured Clinical Interview for DSM-5 (SCID-5) | 0, 6, 12, and 24 months after completion of cognitive behavioral therapy
  Change in the mental disorders diagnosed with the German version of the Structured Clinical Interview for DSM-5
Change in the score on the Beck Depression Inventory-II (BDI-II) | 0, 3, 6, 9, 12, 15, 18, 21, and 24 months after completion of cognitive behavioral therapy
  Change in the score on the German version of the Beck Depression Inventory-II
Change in the score on the WHO (Five) Well-Being Index (WHO-5) | 0, 3, 6, 9, 12, 15, 18, 21, and 24 months after completion of cognitive behavioral therapy
  Change in the score on the German version of the WHO (Five) Well-Being Index
Change in the scores on the Brief-Symptom-Checklist (BSCL) | 0, 3, 6, 9, 12, 15, 18, 21, and 24 months after completion of cognitive behavioral therapy
  Change in the scores on the German short form of the Symptom Checklist-90-Revised
Change in the scores on the Center for Epidemiologic Studies Depression Scale (CES-D) | 0, 3, 6, 9, 12, 15, 18, 21, and 24 months after completion of cognitive behavioral therapy
  Change in the scores on the German version of the Center for Epidemiologic Studies Depression Scale
Change in the scores on the Difficulties in Emotion Regulation Scale (DERS) | 0, 3, 6, 9, 12, 15, 18, 21, and 24 months after completion of cognitive behavioral therapy
  Change in the scores on the German version of the Difficulties in Emotion Regulation Scale
Change in the scores on the Heidelberg Form for Emotion Regulation Strategies (HFERST) | 0, 3, 6, 9, 12, 15, 18, 21, and 24 months after completion of cognitive behavioral therapy
  Change in the scores on the Heidelberg Form for Emotion Regulation Strategies (German questionnaire)

SECONDARY OUTCOMES:
Change in the scores on the Questions on Life Satisfaction (FLZM) | 0, 3, 6, 9, 12, 15, 18, 21, and 24 months after completion of cognitive behavioral therapy
  Change in the scores on the Questions on Life Satisfaction (German Questionnaire)
Change in the scores on the Revised UCLA Loneliness Scale | 0, 3, 6, 9, 12, 15, 18, 21, and 24 months after completion of cognitive behavioral therapy
  Change in the scores on the German version of the Revised UCLA Loneliness Scale
Change in the scores on the Rosenberg's Self-Esteem Scale | 0, 3, 6, 9, 12, 15, 18, 21, and 24 months after completion of cognitive behavioral therapy
  Change in the scores on the revised version of the German adaptation of Rosenberg's Self-Esteem Scale

CONTACTS AND LOCATIONS:
Overall Officials: Verena Zimmermann, M.Sc., Principal Investigator — Department of Clinical Psychology and Psychotherapy, Heidelberg University; Christina Timm, M.Sc., Principal Investigator — Department of Clinical Psychology and Psychotherapy, Heidelberg University; Annemarie Miano, PhD, Principal Investigator — Department of Clinical Psychology and Psychotherapy, Heidelberg University; Sven Barnow, Prof., Principal Investigator — Department of Clinical Psychology and Psychotherapy, Heidelberg University
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Institute of Psychology, Heidelberg University, Heidelberg, Germany

REFERENCES:
- [Background] Beck AT, Steer RA, Brown GK. Beck depression inventory - second edition. Manual. San Antonio, TX: Psychological Corporation, 1996.
- [Background] Beesdo-Baum K, Zaudig M, Wittchen H-U. SCID-5-CV. Strukturiertes klinisches Interview für DSM-5®-Störungen - klinische Version. Deutsche Bearbeitung des structured clinical interview for DSM-5® disorders - clinician version von Michael B. First, Janet B.W. Williams, Rhonda S. Karg, Robert L. Spitzer. Göttingen: Hogrefe Verlag, 2019.
- [Background] Derogatis, LR. SCL-90-R: Administration, scoring, and procedures manual. Baltimore: Clinical Psychometric Research, 1977.
- [Background] Döring N, Bortz J. Psychometrische Einsamkeitsforschung: deutsche Neukonstruktion der UCLA Loneliness Scale. Diagnostica 39(3): 224-239, 1993.
- [Background] Ehring T. Übersetzung und Validierung dreier Instrumente zur Erfassung von Merkmalen der Emotionsregulation [Translation and validation of three instruments for the assessment of characteristics of emotion regulation. In preparation.
- [Background] First MB, Williams JBW, Karg RS, Spitzer RL. Structured clinical interview for DSM-5 disorders, clinician version (SCID-5-CV). Arlington, VA: American Psychiatric Association, 2016.
- [Background] Franke GH. BSCL. Brief-Symptom-Checklist. Göttingen: Hogrefe Verlag, 2012.
- [Background] Gratz KL, Roemer L. Multidimensional assessment of emotion regulation and dysregulation: development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment 26(1): 41-54, 2004.
- [Background] Hautzinger M, Bailer M, Hofmeister D, Keller F. Allgemeine Depressionsskala. 2., überarbeitete und neu normierte Auflage. Göttingen: Hogrefe Verlag, 2012.
- [Background] Hautzinger M, Keller F, Kühner C. BDI-II - Beck Depressions-Inventar - Manual. Frankfurt am Main: Harcourt Test Services, 2006.
- [Background] Henrich G, Herschbach P. Questions on life satisfaction (FLZM) - a short questionnaire for assessing subjective quality of life. European Journal of Psychological Assessment 16(3), 150-159, 2000.
- [Background] Izadpanah S, Barnow S, Neubauer AB, Holl J. Development and Validation of the Heidelberg Form for Emotion Regulation Strategies (HFERST): Factor Structure, Reliability, and Validity. Assessment. 2019 Jul;26(5):880-906. doi: 10.1177/1073191117720283. Epub 2017 Jul 21. PMID 28730850
- [Background] Psychiatric Research Unit, WHO Collaborating Center for Mental Health. WHO (five) well-being index (1998 version). Retrieved from: https://www.psykiatri-regionh.dk/who-5/Documents/WHO5_English.pdf, 1998.
- [Background] Psychiatric Research Unit, WHO Collaborating Center for Mental Health. WHO (fünf) - Fragebogen zum Wohlbefinden (Version 1998). Retrieved from: https://www.psykiatri-regionh.dk/who-5/Documents/WHO5_German.pdf, 1998.
- [Background] Radloff LS. The CES-D scale: a self-report depression scale for research in the general population. Applied Psychological Measurement 3(1): 385-401, 1977.
- [Background] Rosenberg M. Sosciety and the adolescent self-image. Princeton, NJ: Princeton University Press, 1965.
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205
- [Background] von Collani G, Herzberg PY. Eine revidierte Fassung der deutschsprachigen Skala zum Selbstwertgefühl von Rosenberg. Zeitschrift für Differentielle und Diagnostische Psychologie 24(1): 3-7, 2003.